CLINICAL TRIAL: NCT06245525
Title: Palliative Care and Legal Aspects of Treatment Limitation Decisions in ICU: A Survey of Clinicians' Perceptions
Brief Title: Survey on Palliative Care and Law Perception
Acronym: PCLAW
Status: Completed | Type: Observational
Sponsor: University of Athens (Other)
Collaborators: King's College Hospital NHS Trust (Other); University of Southern Denmark (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Spyros D. Mentzelopoulos, Professor of Intensive Care Medicine, National and Kapodistrian University of Athens
Other Study IDs: 606/20/12/2023
Record Dates: First submitted 2024-01-15; First posted 2024-02-07 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: End of Life
Keywords: palliative care; end-of-life legislation; advance directive; do not attempt cardiopulmonary resuscitation; analgesia; sedation; euthanasia; treatment limitation
MeSH Terms: conditions — Death; Agnosia; Suicide, Assisted

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: This is not an interventional study — This is not an interventional study

SUMMARY:
The primary objective of the current survey study is to obtain detailed information about European intensive care unit (ICU) clinicians' awareness of palliative care and relevant, local end-of-life (EoL) legislation.

DETAILED DESCRIPTION:
INTRODUCTION In countries with patient/family autonomy-oriented end-of-life (EOL) legislation, published data indicate variation of healthcare professionals' awareness of the specific legal provisions and/or regulations enabling limitation of life-sustaining treatments. Furthermore, communication difficulties and/or uncertainties about the validity of previously recorded patient preferences (e.g. in the form of advance directives) may result in heterogenous application of pertinent EOL laws/regulations. This may include cases of poor compliance with, or even opposition to new laws.

The absence of accurate and in-depth EOL legal knowledge of clinicians may be associated with perceptions that applicable laws/regulations are either too restrictive or excessively "liberal" for the patient. Furthermore, critical care physicians and/or nurses may lack specific knowledge about palliative care. Accordingly, physicians/nurses may also not be aware of the palliative nature of their everyday practice or have a clear understanding of primary and specialist palliative care.

Given the above-mentioned knowledge gaps of healthcare professionals caring for critically ill patients, the investigators propose to conduct a Europewide, descriptive survey for intensive care unit (ICU) clinicians, primarily aimed at addressing the following questions: 1) "How much of ICU everyday practice is palliative care and how is it practiced?"; and 2) "How do clinicians perceive the medico-legal framework around therapy limitations, patient autonomy and prognostication discussions with patients and families?" In addition, this survey will enable the investigators to comparatively assess the perceived extent of ICU palliative care practice in the presence vs. absence of EOL legislation.

METHODS Study participants and protocol approval The target population of this descriptive, open survey will include ICU physicians and nurses working in at least 100 ICUs across 50 European countries and Israel. Each one of participating ICUs will be represented by one or more healthcare professionals, and the target convenience-sample size will amount to at least 500 respondents (see also below-provided statistical analysis plan). This survey study is part of the European Union-funded Enhancing Palliative Care in ICU (EPIC) project (Proposal number: 101137221; HORIZON-HLTH-2023-DISEASE-03-01). The study protocol has been approved by the Scientific Council of Evaggelismos Hospital, Athens, Greece.

Informed consent and data protection A similar methodology has been recently described. According to the Helsinki declaration, participation in research requires informed consent of the participant. According to Regulation 679/2016 {or General Data Protection regulation (GDPR) of the European Parliament and of the Council, "consent" of the data subject means any freely given, specific, informed and unambiguous indication of the data subject's wishes by which he or she, by a statement or by a clear affirmative action, signifies agreement to the processing of personal data relating to him or her." Participation in and completion of the current survey means that the participant accepts to share their knowledge on palliative care practice, EOL legislation and EOL practice in their country. The estimated time for survey completion is between 30 and 60 min.

The procedure for "pseudonymisation" is detailed below. A set of 20 consecutive random numbers (range, 10-29) will be generated using "Research Randomizer (www.randomizer.org). Each one of the aforementioned numbers will be assigned to a European country (country code) drawn according to alphabetic order from the list of participating countries. Next to the 2 digits of the country code, a one-to-three-digit number will be placed to represent each participant's temporal order of participation relative to other participants from the same country. The country-specific, temporal order of participants will be determined according to the exact time of submission of the completed study questionnaire. This will form the personal, three-to-five digit code for each study participant.

The survey database will be hosted by the CHARITE Berlin Simulation and Training Centre. Data on questionnaire domains will be stored next to the participant's personal code in Microsoft Excel format. This electronic Masterfile will be stored onto the password-protected hard disk of a personal computer. In addition, next to the participant's personal code, investigators will enter the following personal data 1) age; 2) gender; 3) religion; 4 and 5) country and center/city of professional activity; 6) characteristics of the participant's ICU (e.g. general, medical, surgical, etc.); 7) the participant's professional focus (e.g. clinical, research, etc.); and 8 and 9) the participant's professional grade (e.g. consultant, professor, etc.) and ICU experience (in years of work). There will be no collection/recording of participants' names or electronic mail addresses. Therefore, the Masterfile will fulfill the criterion of "pseudonymization." Development and testing of the questionnaire The final version of the questionnaire is presented in the uploaded official and approved version of the current protocol. The questionnaire was developed based on published, relevant literature, investigator consensus and comments collected by preliminary testing; the latter comprised administration of the questionnaire to a total of 30 Danish, British and Greek ICU clinicians (10 from each country). Danish and British clinicians were asked to qualitatively assess the readability and understandability of the survey questions and provide comments for improvement as regards content and clarity. Greek clinicians were asked to first respond to the questionnaire, in order to obtain an estimate of the actual time required for survey completion, and subsequently also provide their comments on content and clarity.

In its finalized form, the survey consists of an introduction and 4 sections. The introduction includes core definitions concerning advance directives and shared decision making, palliative care (https://www.who.int/europe/news-room/fact-sheets/item/palliative-care), treatment limitation, active shortening of the dying process (or euthanasia), and family. The first section aims at collecting data on participant characteristics, including age, gender, religion, location of professional activity (including hospital name), professional focus, grade and experience. The second section includes questions on patient-level, family-level and healthcare-level domains of palliative care, as well as participant-rating (5-point scale) of the importance of domain elements; these elements pertain to physical and psychosocial aspects of care, communication, family support and system-level support. The third section includes questions (and rating by 5-point scale wherever appropriate) about EOL legislation and practices such as applicability of and clinician-compliance with advance directives, treatment limitation (i.e. withholding or withdrawing of life-sustaining treatments), euthanasia, terminal analgesia/sedation, EOL decision-making and family presence during cardiopulmonary resuscitation. Lastly, the fourth section includes 12 questions with two-choice answers (i.e. yes/no) in the context of a recently introduced EOL practice score (with definitions of score subcomponents appended), and an additional 3 general questions about palliative care practice in the participant's ICU.

Website, survey promotion and access to the questionnaire The electronic version of the questionnaire will be set up at a dedicated website using LimeSurvey. Invitation links for this mandatory survey (meaning: all website visitors are expected to fill the survey) will be sent Europe-wide by EPIC partner European Society of Anaesthesiology and Intensive Care (ESAIC) with the use of social media and email channels; ESAIC has approximately 18.000 followers. Additional invitation links will be emailed by the investigators to their networks of research associates; the latter will also be encouraged to share the invitation links with their own networks of colleagues/associates.

Additional protocol features There are no planned incentives for participants. Data collection will be performed once from each participating center, within February 10th to June 30, 2024.

The questionnaire (appended to the current text) will be administered over a total of 22 electronic pages. The items (i.e. subsection questions) per page will range from 1 (open-ended questions) to 12 (multiple-choice questions). Options for responses such as "do not know" are provided for all questions of sections 2 and 3 and question 25.1 of section 4. In addition, adaptive questioning (i.e. "do not know" or "No" responses to the first question of a subsection triggering cancellation of all subsequent questions of that particular subsection) is used from question 15.1 through question 21.1 of section 3; this is aimed at reducing the number of questions in cases of 1) lack of participants' knowledge about whether certain EOL practices are legally allowed; or 2) participant awareness of absence of any preceding/current, local legalization of an EOL practice. In section 4, EOL practice score questions have by original protocol only 2 possible answers, whereas questions 25.2, 25.3 and 25.4 are open ended.

The completeness of participants' responsiveness (i.e. "all survey questions answered") will be checked before questionnaire submission, and participants will be prompted through a "pop-up" dialog box to provide any missing responses, or indicate that they do not wish to respond to a specific question. Furthermore, just prior to questionnaire submission, another "pop-up" dialog box will display a pre-submission prompt to review (and revise if needed) the originally provided responses.

Internet protocol (IP) address data will be used to ensure the uniqueness of survey participants. More specifically, unlimited, repetitive access to the questionnaire will be allowed from an IP address of a client computer until survey submission. However, following submission of the filled questionnaire through an IP address, will result in discontinuation of survey accessibility through that particular IP address.

Due to the use of snowballing dissemination and sharing of invitation links, it will not be possible to calculate the survey response rate. However, survey completion rate will actually be calculated by dividing the total number of submitted questionnaires to the number of first-survey page visitors. Furthermore, questionnaire completeness rate will be calculated by dividing the number of questionnaires without any missing response to the total number of submitted questionnaires. Missing responses will correspond to questions to which participants will have indicated that they do not wish to answer (see also above).

Mutually contradictory responses from participants originating from the same study center, or the same city, or the same country constitute a possibility, especially for the third and fourth section of the survey. For example, two or more participants from the same center/city/country may respond differently as regards the legal bindingness of advance directives. In such cases, mutually contradictory responses will be used to estimate the extent of country-specific variation in the perception of law and/or local palliative care practice.

Outcome Measures Study outcomes are detailed in the dedicated section. Statistical analysis plan Statistical analyses will include 1) descriptive statistics; 2) assessment of distribution normality (by Kolmogorov Smirnov test); 3) assessment of European country-/region-level heterogeneity in the responses; and 4) region-level comparisons of responses.

The investigators expect to determine substantial heterogeneity in the responses, primarily between northern and southern Europe and central and southern Europe, and generally between countries with high vs low palliative care service integration.

High palliative care score will be defined as presence of at least 23 positive responses (out of 35 possible positive responses) to question groups 10 through 14 of survey section 2.

Generalized estimating equations (GEE) models with robust standard errors and exchangeable working correlation structure accounting for the factor center will be applied to examine associations between a high palliative care score, the 9 clinician demographic variables of survey section 1 [with "country" stratified according to "northern, central or southern European region"], and the EOL practice score and/or its subcomponent EOL practice variables listed in question group 24 of survey section 4. The dependent variable in this analysis will be high palliative care score, yes or no. Reference category for region will be "southern Europe". The maximum number of GEE explanatory variables will be 21. Consequently, a target sample size of 500 participants is expected to result in approximately 24 observations (i.e. response data-points) per variable; this exceeds the recommended threshold of 20 observations per variable by 20% and establishes an adequate safety margin, aimed at addressing the possibility of missing responses.

Significance will be set at two-sided P <0.05. Analyses will be conducted using the latest versions of SSPS or R software.

The study questionnaire is included in the uploaded and approved, official version of the study protocol.

Minor modification in the study questionnaire: To ensure data protection, original question No. 5 (in section "clinician demographics") has been changed from "5. Name of hospital/healthcare facility and city of your professional activity (free text)" to "5. Total number of intensive care unit (ICU) beds at your hospital (number)".

ELIGIBILITY:
Inclusion Criteria:

• European and Iraeli intensive care unit physicians or nurses.

Exclusion Criteria:

• Absence of informed consent for study participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Physicians or nurses working in European intensive care units (ICUs), or in ICUs in Israel.
Sampling Method: Non-Probability Sample
Enrollment: 523 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
Clinicians' perceptions of palliative care. | February 1 to July 1 2024.
  The absolute numbers of positive (i.e. yes) responses to question groups 10 through 14 of survey section 2. This will comprise the palliative care score, which ranges from 0 to 24, with greater values indicating a higher quality of palliative care practice.
Clinicians' perceptions of legislation relevant to palliative care. | February 1 to July 1 2024.
  The absolute numbers of positive (i.e. yes) responses to question groups 15 through 23 of section 3. This will comprise the end-of-life legislation score, which ranges from 0 to 49, with greater values indicating higher level of awareness of a comprehensive legal framework.
Clinicians' percreptions of their daily end-of-life and palliative care practice. | February 1 to July 1 2024.
  The absolute numbers of positive (i.e. yes) responses to question groups 24 and 25 of section 4. This will comprise the end-of-life and palliative care practice score, which ranges from 0 to 13, with higher values indicating a higher quality of end-of-life practice.

SECONDARY OUTCOMES:
Clinicians' perceptions of palliative care, in the presence of country end-of-life legislation. | February 1 to July 1 2024.
  The absolute numbers of positive (i.e. yes) responses to question groups 10 through 14, in the presence of a positive response to question 24.12 of section 4. The aforementioned absolute numbers will comprise the palliative care score, which ranges from 0 to 24, with greater values indicating a higher quality of palliative care practice.
Clinicians' perceptions of palliative care, in the absence of country end-of-life legislation. | February 1 to July 1 2024.
  The absolute numbers of positive (i.e. yes) responses to question groups 10 through 14, in the absence of a positive response to question 24.12 of section 4. The aforementioned absolute numbers will comprise the end-of-life legislation score, which ranges from 0 to 49, with greater values indicating higher level of awareness of a comprehensive legal framework.

OTHER OUTCOMES:
Independent predictors of a high palliative care score | February 1 to July 1 2024.
  Generalized estimating equations model-based determination of independent predictors of a high palliative care score. This score ranges from 0 to 24, with greater values indicating a higher quality of palliative care practice. The value of 16 has been specified as the threshold value for a "high" score; this means that palliative care scores of 16 or greater indicate "high-quality" palliative care practice.

CONTACTS AND LOCATIONS:
Overall Officials: Spyros D Mentzelopoulos, MD, PhD, Principal Investigator — National and Kapodistrian University of Athens, Greece; Victoria Metaxa, MD, PhD, Principal Investigator — King's College NHS trust, London; Hanne-Irene Jensen, PhD, CCN, Study Director — Lillebaelt hospital, University of Southern Denmark; Christiane Hartog, MD, PhD, Study Chair — Charite University, Berlin, Germany
Locations (1):
- Evaggelismos General Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Riessen R, Bantlin C, Wiesing U, Haap M. [End-of life decisions in intensive care units. Influence of patient wishes on therapeutic decision making]. Med Klin Intensivmed Notfmed. 2013 Jun;108(5):412-8. doi: 10.1007/s00063-013-0233-3. Epub 2013 Mar 17. German. PMID 23503669
- [Background] Strauss S, Kuppinger D, Hartl WH. [Quality of dying processes after commencement of the German Living Will Act : Experiences of a surgical intensive care unit]. Chirurg. 2017 Mar;88(3):244-250. doi: 10.1007/s00104-016-0345-4. German. PMID 27995297
- [Background] Graw JA, Marsch F, Spies CD, Francis RCE. End-of-Life Decision-Making in Intensive Care Ten Years after a Law on Advance Directives in Germany. Medicina (Kaunas). 2021 Sep 4;57(9):930. doi: 10.3390/medicina57090930. PMID 34577853
- [Background] Doron D, Wexler ID, Shabtai E, Corn BW. Israeli Dying Patient Act: physician knowledge and attitudes. Am J Clin Oncol. 2014 Dec;37(6):597-602. doi: 10.1097/COC.0b013e318295b022. PMID 23660598
- [Background] Boulanger A, Chabal T, Fichaux M, Destandau M, La Piana JM, Auquier P, Baumstarck K, Salas S. Opinions about the new law on end-of-life issues in a sample of french patients receiving palliative care. BMC Palliat Care. 2017 Jan 21;16(1):7. doi: 10.1186/s12904-016-0174-8. PMID 28109272
- [Background] Ciliberti R, Gorini I, Gazzaniga V, De Stefano F, Gulino M. The Italian law on informed consent and advance directives: New rules of conduct for the autonomy of doctors and patients in end-of-life care. J Crit Care. 2018 Dec;48:178-182. doi: 10.1016/j.jcrc.2018.08.039. Epub 2018 Aug 29. PMID 30216936
- [Background] Bonsignore A, Bragazzi NL, Basile C, Pelosi P, Gratarola A, Bonatti G, Patroniti N, Ciliberti R. Development and Validation of a Questionnaire investigating the Knowledge, Attitudes and Practices of Healthcare Workers in the Field of Anesthesiology concerning the Italian Law on Advance Healthcare Directives: a Pilot Study. Acta Biomed. 2021 Sep 2;92(4):e2021092. doi: 10.23750/abm.v92i4.11314. PMID 34487082
- [Background] White B, Willmott L, Cartwright C, Parker MH, Williams G. Knowledge of the law about withholding or withdrawing life-sustaining treatment by intensivists and other specialists. Crit Care Resusc. 2016 Jun;18(2):109-15. PMID 27242109
- [Background] Le Dorze M, Kandelman S, Veber B; SFAR's Ethics Committee. End-of-life care in the French ICU: Impact of Claeys-Leonetti law on decision to withhold or withdraw life-supportive therapy. Anaesth Crit Care Pain Med. 2019 Dec;38(6):569-570. doi: 10.1016/j.accpm.2019.10.013. No abstract available. PMID 31785697
- [Background] Evans N, Bausewein C, Menaca A, Andrew EV, Higginson IJ, Harding R, Pool R, Gysels M; project PRISMA. A critical review of advance directives in Germany: attitudes, use and healthcare professionals' compliance. Patient Educ Couns. 2012 Jun;87(3):277-88. doi: 10.1016/j.pec.2011.10.004. Epub 2011 Nov 23. PMID 22115975
- [Background] Mentzelopoulos SD, Slowther AM, Fritz Z, Sandroni C, Xanthos T, Callaway C, Perkins GD, Newgard C, Ischaki E, Greif R, Kompanje E, Bossaert L. Ethical challenges in resuscitation. Intensive Care Med. 2018 Jun;44(6):703-716. doi: 10.1007/s00134-018-5202-0. Epub 2018 May 10. PMID 29748717
- [Background] Vitale C, de Nonneville A, Fichaux M, Salas S. Medical staff opposition to a deep and continuous palliative sedation request under Claeys-Leonetti law. BMC Palliat Care. 2019 Jan 8;18(1):2. doi: 10.1186/s12904-018-0384-3. PMID 30621684
- [Background] Mercadante S, Gregoretti C, Cortegiani A. Palliative care in intensive care units: why, where, what, who, when, how. BMC Anesthesiol. 2018 Aug 16;18(1):106. doi: 10.1186/s12871-018-0574-9. PMID 30111299
- [Background] Sesma-Mendaza A, Aranguren-Sesma M, Estraviz-Pardo F, Lizarazu-Armendariz E, Goni-Viguria R. Nurses' knowledge about palliative care in a critical care unit. Enferm Intensiva (Engl Ed). 2022 Oct-Dec;33(4):197-205. doi: 10.1016/j.enfie.2021.10.003. Epub 2022 Nov 5. PMID 36347801
- [Background] Mentzelopoulos SD, Couper K, Raffay V, Djakow J, Bossaert L. Evolution of European Resuscitation and End-of-Life Practices from 2015 to 2019: A Survey-Based Comparative Evaluation. J Clin Med. 2022 Jul 11;11(14):4005. doi: 10.3390/jcm11144005. PMID 35887769
- [Background] Mentzelopoulos SD, Couper K, Voorde PV, Druwe P, Blom M, Perkins GD, Lulic I, Djakow J, Raffay V, Lilja G, Bossaert L. European Resuscitation Council Guidelines 2021: Ethics of resuscitation and end of life decisions. Resuscitation. 2021 Apr;161:408-432. doi: 10.1016/j.resuscitation.2021.02.017. Epub 2021 Mar 24. PMID 33773832
- [Background] Sprung CL, Ricou B, Hartog CS, Maia P, Mentzelopoulos SD, Weiss M, Levin PD, Galarza L, de la Guardia V, Schefold JC, Baras M, Joynt GM, Bulow HH, Nakos G, Cerny V, Marsch S, Girbes AR, Ingels C, Miskolci O, Ledoux D, Mullick S, Bocci MG, Gjedsted J, Estebanez B, Nates JL, Lesieur O, Sreedharan R, Giannini AM, Fucinos LC, Danbury CM, Michalsen A, Soliman IW, Estella A, Avidan A. Changes in End-of-Life Practices in European Intensive Care Units From 1999 to 2016. JAMA. 2019 Nov 5;322(17):1692-1704. doi: 10.1001/jama.2019.14608. PMID 31577037
- [Background] Davidson JE, Aslakson RA, Long AC, Puntillo KA, Kross EK, Hart J, Cox CE, Wunsch H, Wickline MA, Nunnally ME, Netzer G, Kentish-Barnes N, Sprung CL, Hartog CS, Coombs M, Gerritsen RT, Hopkins RO, Franck LS, Skrobik Y, Kon AA, Scruth EA, Harvey MA, Lewis-Newby M, White DB, Swoboda SM, Cooke CR, Levy MM, Azoulay E, Curtis JR. Guidelines for Family-Centered Care in the Neonatal, Pediatric, and Adult ICU. Crit Care Med. 2017 Jan;45(1):103-128. doi: 10.1097/CCM.0000000000002169. PMID 27984278
- [Background] Virdun C, Luckett T, Lorenz K, Davidson PM, Phillips J. Dying in the hospital setting: A meta-synthesis identifying the elements of end-of-life care that patients and their families describe as being important. Palliat Med. 2017 Jul;31(7):587-601. doi: 10.1177/0269216316673547. Epub 2016 Dec 8. PMID 27932631
- [Background] Leemans K, Deliens L, Van den Block L, Vander Stichele R, Francke AL, Cohen J. Systematic Quality Monitoring For Specialized Palliative Care Services: Development of a Minimal Set of Quality Indicators for Palliative Care Study (QPAC). Am J Hosp Palliat Care. 2017 Jul;34(6):532-546. doi: 10.1177/1049909116642174. Epub 2016 Apr 7. PMID 27059060
- [Background] Vuong C, Kittelson S, McCullough L, Yingwei Y, Hartjes T. Implementing primary palliative care best practices in critical care with the Care and Communication Bundle. BMJ Open Qual. 2019 Sep 6;8(3):e000513. doi: 10.1136/bmjoq-2018-000513. eCollection 2019. PMID 31544163
- [Background] Mentzelopoulos SD, Bossaert L, Raffay V, Askitopoulou H, Perkins GD, Greif R, Haywood K, Van de Voorde P, Xanthos T. A survey of key opinion leaders on ethical resuscitation practices in 31 European Countries. Resuscitation. 2016 Mar;100:11-7. doi: 10.1016/j.resuscitation.2015.12.010. Epub 2016 Jan 14. PMID 26776899
- [Background] Mentzelopoulos SD, Chen S, Nates JL, Kruser JM, Hartog C, Michalsen A, Efstathiou N, Joynt GM, Lobo S, Avidan A, Sprung CL; End-of-life Practice Score Study Group. Derivation and performance of an end-of-life practice score aimed at interpreting worldwide treatment-limiting decisions in the critically ill. Crit Care. 2022 Apr 13;26(1):106. doi: 10.1186/s13054-022-03971-9. PMID 35418103
- [Background] Avidan A, Sprung CL, Schefold JC, Ricou B, Hartog CS, Nates JL, Jaschinski U, Lobo SM, Joynt GM, Lesieur O, Weiss M, Antonelli M, Bulow HH, Bocci MG, Robertsen A, Anstey MH, Estebanez-Montiel B, Lautrette A, Gruber A, Estella A, Mullick S, Sreedharan R, Michalsen A, Feldman C, Tisljar K, Posch M, Ovu S, Tamowicz B, Demoule A, DeKeyser Ganz F, Pargger H, Noto A, Metnitz P, Zubek L, de la Guardia V, Danbury CM, Szucs O, Protti A, Filipe M, Simpson SQ, Green C, Giannini AM, Soliman IW, Piras C, Caser EB, Hache-Marliere M, Mentzelopoulos SD; ETHICUS-2 Study Group. Variations in end-of-life practices in intensive care units worldwide (Ethicus-2): a prospective observational study. Lancet Respir Med. 2021 Oct;9(10):1101-1110. doi: 10.1016/S2213-2600(21)00261-7. Epub 2021 Aug 6. PMID 34364537
- [Background] Peduzzi P, Concato J, Kemper E, Holford TR, Feinstein AR. A simulation study of the number of events per variable in logistic regression analysis. J Clin Epidemiol. 1996 Dec;49(12):1373-9. doi: 10.1016/s0895-4356(96)00236-3. PMID 8970487

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-15): https://cdn.clinicaltrials.gov/large-docs/25/NCT06245525/Prot_SAP_000.pdf